CLINICAL TRIAL: NCT06978400
Title: Non-randomised, Multicentre, Prospective, Single-arm, Phase II Study of the Efficacy and Toxicity of a Combination of FOLFOX With Dabrafenib and Cetuximab/Panitumumab in the First Line of Therapy of Patients With Metastatic BRAF V600E- Mutated MSS Colorectal Cancer
Brief Title: A Study of Dabrafenib Plus Cetuximab/Panitumumab With FOLFOX in the First Line of Therapy in People With Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Collaborators: City Clinical Oncology Hospital No 1 (Other Government); Moscow City Oncology Hospital No. 62 (Other Government); The Loginov MCSC MHD (Unknown); MMCC Kommunarka MHD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05202500303
Record Dates: First submitted 2025-05-03; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Neoplasms
Keywords: metastatic colorectal cancer; BRAF V600E- mutated; first line; MSS; treatment
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms | interventions — dabrafenib; Cetuximab; Panitumumab

STUDY DESIGN:
Intervention Model Description: * Drug: Dabrafenib
  * Drug: Cetuximab
  * Drug: Рanitumumab
  * Drug: Oxaliplatin
  * Drug: Irinotecan
  * Drug: Leucovorin
  * Drug: 5-FU
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mFOLFOX6 + dabrafenib and cetuximab or panitumumab in the first line of therapy (Experimental): mFOLFOX6 + dabrafenib and cetuximab or panitumumab in the first line of therapy Dabrafenib 150 mg twice orally daily Cetuximab 500 mg/m2 (120-minute IV infusion) every two weeks or Panitumumab 6 mg/kg (60-minute IV infusion) every two weeks Oxaliplatin 85 mg/m2 (120-minute IV infusion) every two weeks, Сalcium folinate 400 mg/m2 (120-minute IV infusion) every two weeks 5-FU 400 mg/m2 IV bolus, then 5-FU 2400 mg/m2 continuous IV infusion over 46-48 hours every two weeks.
  In the first-line setting, 8 courses are administered, and if disease control is achieved, dabrafenib, cetuximab or panitumumab therapy is continued until disease progression or intolerable toxicity.
  Interventions: Drug: mFOLFOX6 + dabrafenib and cetuximab or panitumumab in the first line of therapy

INTERVENTIONS:
Drug: mFOLFOX6 + dabrafenib and cetuximab or panitumumab in the first line of therapy — Dabrafenib 150 mg twice orally daily Cetuximab 500 mg/m2 (120-minute IV infusion) every two weeks or Panitumumab 6 mg/kg (60-minute IV infusion) every two weeks Oxaliplatin 85 mg/m2 (120-minute IV infusion) every two weeks, Сalcium folinate 400 mg/m2 (120-minute IV infusion) every two weeks 5-FU 400 mg/m2 IV bolus, then 5-FU 2400 mg/m2 continuous IV infusion over 46-48 hours every two weeks.

SUMMARY:
The purpose of this study is to evaluate the efficacy and toxicity of FOLFOX regimen with dabrafenib and cetuximab/panitumumab in the first line of therapy for the potential treatment of colorectal cancer that: has a metastatic, inoperable; has a mutation in the BRAF gene and MSS.

Participants in this study will receive one of the following study treatments:

These participants will receive FOLFOX regimen with dabrafenib and cetuximab or panitumumab in the first line of therapy This study is currently enrolling participants who will receive either FOLFOX regimen with dabrafenib and cetuximab or panitumumab in the first line of therapy.

The study team will monitor how each participant responds to the study treatment for up to about 3 years.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the efficacy and toxicity of first-line FOLFOX with dabrafenib and cetuximab or panitumumab in patients with previously untreated metastatic inoperable colorectal cancer who have MSS and BRAF mutation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal adenocarcinoma that contains MSS and BRAF V600E mutation
* Metastatic inoperable colorectal cancer
* Adequate function of hematopoiesis and basic indicators of internal organs
* Has measurable or evaluable disease according to Response Evaluation Criteria In Solid Tumors (RECIST v1.1).
* Lacking antitumor systemic treatment for colorectal cancer.
* Patients with progression after adjuvant chemotherapy may be included if progression is recorded no earlier than 12 months after the last course of chemotherapy.
* The primary tumor is removed or asymptomatic.
* Absence of grade 2 or higher neuropathy.
* Absence of tumor MSI or dMMR.
* ECOG PS 0-2

Exclusion Criteria:

* Participants having more than 2 lines of treatment (a progression of disease within 12 months of the completion of adjuvant and/or perioperative chemotherapy with oxaliplatin and fluoropyrimidines is acceptable).
* Presence of any other malignancy, except radically treated basal cell carcinoma, cervical cancer in situ, currently or within 5 years prior to enrolment.
* Pregnant and breastfeeding women.
* Male and female patients with preserved reproductive potential who refused to use adequate contraception throughout the study.
* HIV-infected patients.
* Patients with a life expectancy of less than 3 months.
* The presence of a disease or condition that, in the opinion of the investigator, prevents the patient from participating in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-11-10 (Estimated); Study Completion 2028-07-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | assessed at 8 and 16 weeks
  From date of enrollment until the date of first documented objective response

SECONDARY OUTCOMES:
Progression-free survival | assessed up to 24 months
  From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first
Time to objective response | assessed up to 12 months
  Time from start of treatment to objective response to treatment
Overall survival | assessed up to 36 months
  From the time of enrolment until the death from any cause

OTHER OUTCOMES:
Duration of response | assessed up to 12 months
  Calculated from achieving objective response to progression or death from any cause
Disease control rate | through study completion, an average of 1 year
  Percentage of patients who achieved a complete response, partial response or disease stabilisation
Incidence of adverse events | through study completion, an average of 1 year
  Proportion of patients with adverse events out of all patients (NCI CTCAE 5.0)
Incidence of adverse events grade 3-4 | through study completion, an average of 1 year
  Proportion of patients with adverse events grade 3-4 out of all patients (NCI CTCAE 5.0)
Frequency of dose reductions and drug withdrawals | through study completion, an average of 1 year
  Proportion of patients with dose reductions and drug withdrawals in the total number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Fedyanin MD, Principal Investigator — Blokhin's Russian Cancer Research Center
Locations (1):
- Blokhin's Russian Cancer Research Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No